CLINICAL TRIAL: NCT04237948
Title: tDCS Plus Physical Therapy for Progressive Supranuclear Palsy: a Double Blind Randomized Sham-controlled Study With Wearing Sensors Technology
Brief Title: tDCS Plus Physical Therapy for Progressive Supranuclear Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Europea di Ricerca Biomedica Ferb Onlus (Other)
Collaborators: Università degli Studi di Brescia (Other); University of Kiel (Other)
Responsible Party: Principal Investigator, Andrea Pilotto, Parkinson's disease Rehabilitation Centre, Fondazione Europea di Ricerca Biomedica Ferb Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/02
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Progressive Supranuclear Palsy; Parkinsonism; Parkinsonian Disorders
Keywords: tDCS; transcranial direct current stimulation; falls; postural instability; wearing sensors; physical therapy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinsonian Disorders | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two randomized double blind groups will be evaluated. Both group will undergo physical rehabilitation. The real arm group will undergo real cerebellar tDCS while the placebo-arm will undergo a sham stimulation
Who Masked: Participant, Investigator
Masking Description: The patient and the examiner who did the ratings were blind to the type of tDCS delivered, which was applied by another blinded experimenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy plus REAL tDCS (Active Comparator): Patients will be undergo a rehabilitation treatment during hospitalization consisting in 60 minutes of physical rehabilitation for 4 weeks.
  Real Cerebellar tDCS will be applied for 10 days of time.
  Interventions: Device: transcranial direct current stimulation (tDCS); Behavioral: Physical therapy
- physical therapy plus SHAM tDCS (Placebo Comparator): Patients will be undergo a rehabilitation treatment during hospitalization consisting in 60 minutes of physical rehabilitation for 4 weeks.
  Sham Cerebellar tDCS will be applied for 10 days of time.
  Interventions: Behavioral: Physical therapy

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — cerebellar tDCS consists in the application of a low intensity (1-2 mA) steady current through a surface scalp electrode over the cerebellum
  Arms: physical therapy plus REAL tDCS
Behavioral: Physical therapy — Hospitalized patients will undergo a 60 minutes physical treatment improving gait and postural instability for four weeks of time

SUMMARY:
Objective of the study:

To test the efficacy of cerebellar transcranial direct current stimulation (tDCS) associated with physical rehabilitation on postural instability and falls in progressive supranuclear palsy using a double-blind design and wearing sensors technology

Design:

Twenty probable PSP patients with no dementia and still able to walk will be recruited for a randomized double-blind sham-controlled study. Each patient will be hospitalized for a four week physical rehabilitation. In the real-arm, the patients will undergo a ten cerebellar tDCS stimulations while the placebo arm will undergo sham stimulation.

Each patient will be evaluated before and after stimulation by PSP-rating scale (PSP-RS), cognitive tests and a battery of gait and movement tests using wearing sensors technology.

DETAILED DESCRIPTION:
Background:

There are no medical effective treatments for progressive supranuclear palsy (PSP). Imaging, neurophysiology and pathology studies suggested cerebellum as possible target of brain stimulation for postural instability using tDCS stimulation

Objective of the study:

To test the efficacy of cerebellar transcranial direct current stimulation (tDCS) associated with physical rehabilitation on postural instability and falls in progressive supranuclear palsy using a double-blind design and wearing sensors technology

Design:

Twenty probable PSP patients with no dementia and still able to walk will be recruited for a randomized double-blind sham-controlled study. Each patient will be hospitalized for a four week physical rehabilitation. In the real-arm, the patients will undergo a 10 days cerebellar tDCS stimulation while the placebo arm will undergo sham stimulation.

cerebellar tDCS consists in the application of a low intensity (1-2 mA) steady current through a surface scalp electrode over the cerebellum for ten days.

Each patient will be evaluated before and after stimulation by berg balance tests (BBS), Tinetti scale, PSP-rating scale (PSP-RS), cognitive assessment and a battery of gait and movement tests using wearing sensors technology.

Sensors assessment:

The following parameters will be evaluated before and after stimulation (real vs sham): The parameter for postural instability defined are:

i) TIME, defined as time without falling ii) The parameter "surface", defined as the sway area iii) Velocity describes the mean velocity of the compensatory movements given in mm/s. iv) Acceleration described as root mean square (RMS), v) Jerk, the time derivate of acceleration, quantifies smoothness of the compensatory movements given in mG/s.

The parameter for gait and turning evaluation during normal walk and timed up and go, defined are: i) stealth length ii) step variability iii) step phases duration iv) gait speed v) turning velocity

ELIGIBILITY:
Inclusion Criteria:

probable PSP diagnosis ability to stand alone without support for at least 5 seconds ability to walk without aid for at least three meters

Exclusion Criteria:

dementia or behavioral alterations contraindications of stimulation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
PSP rating scale (PSP-RS) | Changes from Baseline to immediately after stimulation and after 3 months
  Assessment of postural instability and disability of patients (scores ranging from 0 to 100, lower scores indicate less disability)
Falls | Number of falls recorded starting from immediately after stimulation until 3 months after the end of stimulation
  Number of falls will be recorded using a diary
Cognitive testing | Changes from Baseline to immediately after stimulation
  Total Z-scores of cognitive assessment (including eight tests assessing memory, executive function, attention and visual-spatial function)
Static Balance- area of sway | Changes from Baseline to immediately after stimulation
  The area of sway during the postural instability tasks will be assessed (unit of measure mm2)

SECONDARY OUTCOMES:
Tinetti Balance test (TBT) | Changes from Baseline to immediately after stimulation and after 3 months
  Assessment of postural instability (0-28, higher scores indicate better performances)
Static Balance: wearable sensor analyses - velocity | Changes from Baseline to immediately after stimulation
  the velocity of sway will be assessed during the postural instability tasks (unit of measure (mm/s)
Gait speed | Changes from Baseline to immediately after stimulation
  The speed of gait will be assessed in one minute of normal and dual-task walking
Turning speed | Changes from Baseline to immediately after stimulation
  The velocity of turning will be assessed in timed up and go tests
Activity of daily living | Changes from Baseline to immediately after stimulation
  the dependence of patient in ADL will be assessed with the help of caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilotto, MD, Principal Investigator — FERB onlus
Locations (1):
- Parkinson's disease Rehabilitation Centre - FERB ONLUS, Trescore Balneario, Italy

IPD SHARING:
Plan to Share IPD: Yes
The whole project will be published in medical journal
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In the publication, within the next year
Access Criteria: on-line free access